CLINICAL TRIAL: NCT03242434
Title: A Prospective, Longitudinal Study to Investigate the Effect of Thermal Injury on Intestinal Permeability and Systemic Inflammation (HESTIA)
Brief Title: Investigation of Thermal Injury on Intestinal Permeability in Both Thermal Injury and Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This trial was supporting the development of an asset which was terminated, thus the data from the study were no longer required.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 206243
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Burns
Keywords: Mannitol; Intestinal permeability; Thermal injury; HESTIA; Sucralose; Lactulose
MeSH Terms: conditions — Burns | interventions — Lactulose; trichlorosucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy controls (Other): Approximately 15 healthy participants of age 18 years or above will be included in the study and will receive STM intermittently via oral route. The total duration of study for healthy participants will be approximately 2 weeks.
  Interventions: Other: Lactulose and Mannitol solution; Other: Sucralose
- Thermal injury participants (Other): Approximately 25 thermally injured participants having TBSA more than or equal to 15 percent and who are co-consented to the SIFTI-2 and HESTIA studies will be included in the study and will receive STM intermittently via oral route. The total duration of study for thermal injury participants will be approximately 6 months.
  Interventions: Other: Lactulose and Mannitol solution; Other: Sucralose

INTERVENTIONS:
Other: Lactulose and Mannitol solution — Participants will receive 100 milliliter (mL) oral solution of Lactulose [5 grams (g)]/ Mannitol (2g), a non-investigational medicinal product, by oral route to measure intestinal permeability.
Other: Sucralose — Participants will receive 3 capsules of Sucralose (2g), a non-investigational medicinal product, by oral route to measure intestinal permeability.

SUMMARY:
This longitudinal, prospective study aims to establish the magnitude and time course of changes in intestinal permeability; establish the optimal method for assessment of intestinal permeability in thermally injured participants: describe the participant population most likely to benefit from a new medicinal product which could prevent changes in intestinal permeability; and improve our understanding of the links between intestinal damage, changes in the gut microbiome and microbial translocation to the systemic circulation following thermal injury. The key factors of interest in this study are to understand the impact of thermal injury on intestinal permeability in thermally injured participants compared to healthy participants; and to understand the changes in intestinal permeability over time. Approximately 15 eligible healthy participants and 25 thermally injury participants will be included. The sugar test material (STM) comprises of Lactulose, Mannitol and Sucralose and will be intermittently administered enterally to all the participants. The full duration of the study for healthy participants will be approximately two weeks and 6 months for thermally injured participants. In order to enter this study thermally injured participants will be required to co-enroll in this study and an allied study entitled: A Multi-center, Prospective Study to Examine the Relationship between Neutrophil Function and Sepsis in Adults and Children with Severe Thermal Injury (SIFTI-2). (reference number IRAS ID: 200366).

ELIGIBILITY:
Inclusion Criteria:

For Healthy participants:

* Males or females must be greater than or equal to 18 years of age at the time of signing informed consent.
* Participants who are healthy as determined by the investigator following medical evaluation including medical history, physical examination, and laboratory tests.
* A female participant is eligible to participate if she is not pregnant (negative pregnancy testing at screening or Day 1 as needed) and not breastfeeding.
* Capable of giving signed informed consent.

For Thermally injured participants:

* Participants must be greater than or equal to 18 years of age.
* Participants who have sustained a burn (thermal injury) with a Total Burn Surface Area (TBSA) greater than or equal to 15 percent.
* Admission to the burn center (study site) less than or equal to 24 hours following injury.
* Able to take enteral fluids either orally or via a nasogastric tube (depends on facial burn damage).
* A female participant is eligible to participate if she is not pregnant (negative pregnancy testing at study entry) and not breastfeeding.

Exclusion Criteria

For Healthy participants:

* Healthy participants are excluded from this study if they are receiving anti-coagulation therapy.
* Pregnancy or breastfeeding.
* A body mass index greater than 34 kilogram per meter square (kg/m^2).
* An active history of alcohol dependency.
* History of sensitivity to any of the STM, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator and/or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody and confirmatory Hepatitis C Polymerase Chain Reaction (PCR) result within 3 months of screening.
* A positive pre-study urine drug/alcohol screen.
* A positive test for Human Immuno-deficiency Virus (HIV) antibody.
* Participants unable to swallow large capsules (the capsules will be shown to participants at screening).
* Galactosaemia or severe lactose intolerance.
* Use of an antibiotic 2 weeks prior to study start (administration of the STM).
* Gastroenteritis in the 2 weeks prior to study start (administration of the STM).

For thermally injured participants:

* Chemical or electrical burn.
* Multiple traumatic injuries with an Injury Severity Score (ISS) more than or equal to 16.
* Participants received substantial undocumented management prior to arrival at the study site (burn center) e.g. from paramedics or in a local accident and emergency department.
* Systemic corticoidsteroid use.
* Intravenous (IV) Mannitol use.
* HIV infection.
* Viral Hepatitis B or C infection.
* Gastrointestinal disease (e.g. inflammatory bowel disease) which may affect intestinal permeability.
* Previous bowel resection (e.g. hemicolectomy, small bowel resection).
* Galactosaemia or severe lactose intolerance.
* Bowel obstruction.
* Renal dysfunction requiring renal replacement therapy (end-stage renal failure prior to thermal injury).
* Active autoimmune disease and receiving immunomodulatory therapy e.g. rheumatoid arthritis anti-Tumor Necrosis Factor (TNF).
* Active chemotherapy for cancers or immunoremittive therapies (prednisolone, Adalimumab) within 60 days of thermal injury.
* Premorbid conditions of malignancy currently under treatment.
* Previous bilateral lower extremity amputation.
* Decision not to treat the participant due to futility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a longitudinal study which involved healthy participants and participants who had sustained a thermal injury. The study was conducted in United Kingdom. This study was terminated early prior to the full sample size being achieved as the development of the formulation was terminated.
Pre-assignment Details: A total 23 participants were screened for study of which 5 participants were screen failure and 18 participants were enrolled in the study.
Groups:
- Healthy Participants: Healthy participants were invited to donate a blood sample for biomarker measurement on day one. They were also requested to undergo measurements of intestinal permeability by taking a 100 milliliter (mL) solution of lactulose (5 gram [g]) and mannitol (2g) along with 3 capsules (2g) of sucralose on days 1, 8 and 15 followed by a 24 hour urine collection.
- Thermal Injury Participants: Participants were invited to undergo measurements of intestinal permeability by taking a 100 mL solution of lactulose (5 g) and mannitol (2g) along with 3 capsules (2g) of sucralose on days 1,3,5,7,9,11 and 13.
Period: Overall Study
Arm/Group | Healthy Participants | Thermal Injury Participants
Started | 15 | 3
Completed | 15 | 1
Not Completed | 0 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Population: One participant from healthy participants was excluded due to protocol deviation.
Groups:
- Thermally Injured Participants: Participants were invited to undergo measurements of intestinal permeability by taking a 100 mL solution of lactulose (5 g) and mannitol (2g) along with 3 capsules (2g) of sucralose on days 1,3,5,7,9,11 and 13.
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Thermally Injured Participants | Total
Number analyzed (Participants) | 14 | 3 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] — Evaluable Population.
  Years | 41.4 (9.43) | 52.0 (21.00) | 43.3 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants] — Evaluable Population
  Participants
    Female | 8 | 1 | 9
    Male | 6 | 2 | 8
Race/Ethnicity, Customized [Number; unit: Count of Participants] — Evaluable Population
  Count of Participants
    Central/South Asian Heritage | 1 | 0 | 1
    White | 13 | 2 | 15
    Black or African American | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From 0 to 5 Hours, and 0 to 24 Hours in the Ratio of Lactulose/Mannitol on Day 1
Description: Urine samples were collected at indicated time-points to determine the impact of thermal injury on the magnitude of small intestine permeability following the injury. As, L/M does not get metabolized, it gets filtered in the kidney and excreted in the urine. The impact of injury in thermal injury participants was compared with healthy participants using L/M ratio in urine.
Time Frame: 0 to 5 hours and 0 to 24 hours on Day 1
Population: Evaluable Population included of all participants in the safety population excluding any healthy volunteers that received any concomitant medication or food and drink containing Sugar Test Material (STM) as identified by review of the protocol deviation. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Thermally Injured Participants: Participants were invited undergo measurements of intestinal permeability by taking a 100 mL solution of lactulose (5 g) and mannitol (2g) along with 3 capsules (2g) of sucralose on days 1,3,5,7,9,11 and 13.
Arm/Group | Healthy Participants | Thermally Injured Participants
Number analyzed (Participants) | 7 | 3
Ratio
  Day 1, 0 to 5 hours | 0.0078 (0.00102) | 0.0415 (0.06243)
  Day 1, 0 to 24 hours | 0.0093 (0.00409) | 0.0296 (0.04031)

2. Primary Outcome: Change From 0 to 5 Hours, and 0 to 24 Hours in the Ratio of Lactulose/Mannitol Over Time for Healthy Participants
Description: Urine samples were collected at indicated time-points to determine the impact of thermal injury on the magnitude of small intestine permeability following the injury. As, L/M does not get metabolized, it gets filtered in the kidney and excreted in the urine. Baseline value was considered as Day 1 for both the groups. Change from Baseline is equal to post-Baseline visit value minus Baseline value.
Time Frame: 0 to 5 hours and 0 to 24 hours on Day 8 and Day 15
Population: Evaluable Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Healthy Participants
Number analyzed (Participants) | 5
Ratio
  Day 8 (0-5 hours) | 0.0132 (0.020600)
  Day 15 (0-5 hours) | 0.0016 (0.00548)
  Day 8 (0-24 hours) | 0.0092 (0.01304)
  Day 15 (0-24 hours) | 0.0090 (0.00698)

3. Primary Outcome: Change From 0 to 5 Hours, and 0 to 24 Hours in the Ratio of Lactulose/Mannitol Over Time for Thermal Injury Participants
Description: as for outcome 2
Time Frame: 0 to 5 hours on Days 3, 5, 7, 11, 13 and 0 to 24 hours on Days 3, 5, 7, 9, 11 and 13
Population: Evaluable Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Thermally Injured Participants
Number analyzed (Participants) | 3
Ratio
  Day 3, (0-5 hours), n= 3 | -0.0037 (0.09936)
  Day 5, (0-5 hours), n= 3 | -0.0213 (0.08213)
  Day 7, (0-5 hours), n= 2: number analyzed (Participants) | 2
  Day 7, (0-5 hours), n= 2 | 0.0566 (0.07509)
  Day 11, (0-5 hours), n= 1: number analyzed (Participants) | 1
  Day 11, (0-5 hours), n= 1 | -0.1044 (NA) — NA indicates data was not available as standard deviation could not be calculated for one participant.
  Day 13, (0-5 hours), n= 1: number analyzed (Participants) | 1
  Day 13, (0-5 hours), n= 1 | -0.0043 (NA) — NA indicates data was not available as standard deviation could not be calculated for one participant.
  Day 3, (0-24 hours), n= 3 | 0.0111 (0.09085)
  Day 5, (0-24 hours), n= 3 | -0.0046 (0.06456)
  Day 7, (0-24 hours), n= 2: number analyzed (Participants) | 2
  Day 7, (0-24 hours), n= 2 | 0.0178 (0.02640)
  Day 9, (0-24 hours), n= 2: number analyzed (Participants) | 2
  Day 9, (0-24 hours), n= 2 | -0.0327 (0.05953)
  Day 11, (0-24 hours), n= 2: number analyzed (Participants) | 2
  Day 11, (0-24 hours), n= 2 | -0.0218 (0.05846)
  Day 13, (0-24 hours), n= 1: number analyzed (Participants) | 1
  Day 13, (0-24 hours), n= 1 | -0.0634 (NA) — NA indicates data was not available as standard deviation could not be calculated for one participant.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAE) and Non-SAE were collected from Day 1 up to 6 months for thermal injury participants and SAE and Non-SAE were collected from Day 1 up to Day 15 for healthy participants. Safety Population comprised of all participants who received at least one dose of STM and have at least one post-dose safety assessment.
Description: Death is typically associated with the disease under study and were not reported as SAEs but instead were recorded drug related events (DREs). In thermally injured participants DREs are common and can be serious/life threatening: Deterioration of condition; Death (may be expected in burns of a large surface area); Prolongation of hospital stay; Persistent or significant disability or incapacity.
Arm/Group | Healthy Participants | Thermally Injured Participants
All-Cause Mortality (participants affected / at risk) | 0/15 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/3
Other Adverse Events (participants affected / at risk) | 5/15 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=15) | Thermally Injured Participants (N=3)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03242434/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT03242434/SAP_001.pdf